CLINICAL TRIAL: NCT02635620
Title: Changes in Lung Function Parameters, Bronchial Reactivity, State of Health and Smoking Behaviour Associated With Changing From Conventional Smoking to Electronic Cigarettes
Brief Title: Changes in Psychological and Somatic Parameters Associated With Changing From Smoking to E-cigarettes
Acronym: EQualLife
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Oliver Pogarell, Prof. Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: EQualLife
Record Dates: First submitted 2015-12-11; First posted 2015-12-21 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Exposure to Electronic Cigarettes
Keywords: e-cigarette, electronic cigarette, lung function
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- e-cigarette group: Probands are smokers who intend to start vaping for the first time. The probands are recruited in e-cigarette shops. It is aimed to include 60 persons who start vaping. A baseline visit at the beginning will measure conventional lung function parameters, mannitol provocation, FeNO and exhaled CO. The measurement will be repeated after 3 months to evaluate changes in these parameters. In addition there will be questionnaires concerning smoking/vaping behaviour and health status at the beginning and after 1, 2 and 3 months.
- smoking cessation group: Probands are smokers who intend to quit smoking within a clinical conducted smoking cessation program. It is aimed to include 20 persons who stop smoking. Like in the e-cigarette group, a baseline visit at the beginning will measure conventional lung function parameters, mannitol provocation, FeNO and exhaled CO. The measurement will be repeated after 3 months to evaluate changes in these parameters. In addition there will be questionnaires concerning smoking behaviour and health status at the beginning and after 1, 2 and 3 months.

SUMMARY:
The purpose of this study is to investigate whether changing from conventional smoking to electronic cigarettes causes changes in conventional lung function parameters, bronchial reactivity, fractional exhaled nitric oxide (FeNO), Carbon monoxide (CO), health effects and smoking behaviour.

DETAILED DESCRIPTION:
STUDY BACKGROUND / RATIONALE / PURPOSE:

There is still little known about the health effects by vaping electronic cigarettes. Some former studies investigated the short term effects of vaping regarding lung function, respiratory resistance and FeNO (fractional exhaled nitric oxide). Flouris et al., 2013 did not found significant short term effects on conventional lung function parameters. Vardavas et al., 2012 also found no short term effects on conventional lung function parameters, but an increase of respiratory resistance and a decrease of FeNO. In contrast, Schober et al., 2014 observed an increase of FeNO after vaping electronic cigarettes.

Experimental studies have shown, that electronic cigarettes induce an inflammatory process in epithelial cells (Lerner et al., 2015; Wu, Jiang, Minor, and Chu, 2014). Lim and Kim, 2014 investigated the effects of e-liquids on the airway reactivity and inflammation on allergic sensitized mice. Reactivity and inflammation got worse.

Long term data is still missing. For this purpose we want to investigate lung function, airway reactivity, health status and smoking/vaping behaviour in smokers at the time they intend to start vaping and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* smoking ≥ 5 years
* smoking ≥ 10 cigarettes per day
* no intention to stop smoking within the last 3 months
* using e-cigarettes with nicotine
* no infection of airways at the time of measurements
* e-cigarette group: intending to use e-cigarettes
* control group: smoking cessation in the framework of a clinical conducted program

Exclusion Criteria:

* pregnancy or breastfeeding
* not speaking German
* known allergy
* acute psychiatric diseases, suicidal tendency
* drug/substance/alcohol abuse
* severe internal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of smokers who want to start using electronic cigarettes.
  Control group contains smokers who stop smoking in the framework of a clinical conducted program.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
lung function | 3 months
  Tiffeneau-Index
quality of life | 3 months
  WHO quality of life - questionary
respiratory tract inflammation activity | 3 months
  FeNO (exhaled nitric oxide)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Rüther, Dr., Principal Investigator — LMU - Munich
Locations (1):
- Klinik für Psychiatrie und Psychotherapie - LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flouris AD, Chorti MS, Poulianiti KP, Jamurtas AZ, Kostikas K, Tzatzarakis MN, Wallace Hayes A, Tsatsakis AM, Koutedakis Y. Acute impact of active and passive electronic cigarette smoking on serum cotinine and lung function. Inhal Toxicol. 2013 Feb;25(2):91-101. doi: 10.3109/08958378.2012.758197. PMID 23363041
- [Background] Schober W, Szendrei K, Matzen W, Osiander-Fuchs H, Heitmann D, Schettgen T, Jorres RA, Fromme H. Use of electronic cigarettes (e-cigarettes) impairs indoor air quality and increases FeNO levels of e-cigarette consumers. Int J Hyg Environ Health. 2014 Jul;217(6):628-37. doi: 10.1016/j.ijheh.2013.11.003. Epub 2013 Dec 6. PMID 24373737
- [Background] Lerner CA, Sundar IK, Yao H, Gerloff J, Ossip DJ, McIntosh S, Robinson R, Rahman I. Vapors produced by electronic cigarettes and e-juices with flavorings induce toxicity, oxidative stress, and inflammatory response in lung epithelial cells and in mouse lung. PLoS One. 2015 Feb 6;10(2):e0116732. doi: 10.1371/journal.pone.0116732. eCollection 2015. PMID 25658421
- [Background] Lim HB, Kim SH. Inhallation of e-Cigarette Cartridge Solution Aggravates Allergen-induced Airway Inflammation and Hyper-responsiveness in Mice. Toxicol Res. 2014 Mar;30(1):13-8. doi: 10.5487/TR.2014.30.1.013. PMID 24795794
- [Background] Wu Q, Jiang D, Minor M, Chu HW. Electronic cigarette liquid increases inflammation and virus infection in primary human airway epithelial cells. PLoS One. 2014 Sep 22;9(9):e108342. doi: 10.1371/journal.pone.0108342. eCollection 2014. PMID 25244293
- [Background] Vardavas CI, Anagnostopoulos N, Kougias M, Evangelopoulou V, Connolly GN, Behrakis PK. Short-term pulmonary effects of using an electronic cigarette: impact on respiratory flow resistance, impedance, and exhaled nitric oxide. Chest. 2012 Jun;141(6):1400-1406. doi: 10.1378/chest.11-2443. Epub 2011 Dec 22. PMID 22194587